CLINICAL TRIAL: NCT04180488
Title: Master Protocol of Three Randomized, Double-blind, Placebo Controlled, Multi-center, Parallel-group Studies of Dupilumab in Patients With Chronic Spontaneous Urticaria (CSU) Who Remain Symptomatic Despite the Use of H1 Antihistamine Treatment in Patients naïve to Omalizumab and in Patients Who Are Intolerant or Incomplete Responders to Omalizumab
Brief Title: Dupilumab for the Treatment of Chronic Spontaneous Urticaria in Patients Who Remain Symptomatic Despite the Use of H1 Antihistamine and Who Are naïve to, Intolerant of, or Incomplete Responders to Omalizumab (LIBERTY-CSU CUPID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC16461; U1111-1241-8208 (Registry Identifier: ICTRP); 2019-003775-19 (EudraCT Number)
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Study A Dupilumab (Experimental): Participants who were omalizumab naïve received dupilumab for 24 weeks as follows:
  * 300 milligrams (mg) SC injection every 2 weeks (q2w) for adults and those adolescents who weighed >=60 kilograms (kg) at screening starting from Week 2 following a loading dose of 600 mg (2×300 mg injections) on Day 1,
  * 200 mg SC injection q2w for adolescents who weighed <60 kg and children (>=6 to <12 years of age) who weighed >=30 kg at screening starting from Week 2 following a loading dose of 400 mg (2×200 mg injections) on Day 1 and
  * 300 mg SC injection every 4 weeks (q4w) for children (>=6 to <12 years of age) who weighed <30 kg and >=15 kg at screening starting from Week 4 following a loading dose of 600 mg (2×300 mg injections) on Day 1.
  Interventions: Drug: Dupilumab SAR231893; Drug: non sedating H1-antihistamine
- Study A Placebo (Placebo Comparator): Participants who were omalizumab naïve received placebo matched to dupilumab as subcutaneous (SC) injection including loading dose from Day 1 up to 24 weeks.
  Interventions: Drug: Placebo; Drug: non sedating H1-antihistamine
- Study B Dupilumab (Experimental): Participants who were intolerant or incomplete responders to omalizumab received dupilumab for 24 weeks as follows:
  * 300 mg SC injection q2w for adults and those adolescents weighing >=60 kg at screening starting from Week 2 following a loading dose of 600 mg (2×300 mg injections) on Day 1 or
  * 200 mg SC injection q2w for adolescents weighing <60 kg at screening starting from Week 2 following a loading dose of 400 mg (2×200 mg injections) on Day 1.
  Interventions: Drug: Dupilumab SAR231893; Drug: non sedating H1-antihistamine
- Study B Placebo (Placebo Comparator): Participants who were intolerant or incomplete responders to omalizumab received placebo matched to dupilumab as SC injection including loading dose from Day 1 up to 24 weeks.
  Interventions: Drug: Placebo; Drug: non sedating H1-antihistamine
- Study C Dupilumab (Experimental): Participants who were omalizumab naïve received dupilumab for 24 weeks as follows:
  * 300 mg SC injection q2w for adults and those adolescents who weighed >=60 kg at screening starting from Week 2 following a loading dose of 600 mg (2×300 mg injections) on Day 1,
  * 200 mg SC injection q2w for adolescents who weighed <60 kg and children (>=6 to <12 years of age) who weighed >=30 kg at screening starting from Week 2 following a loading dose of 400 mg (2×200 mg injections) on Day 1 and
  * 300 mg SC injection q4w for children (>=6 to <12 years of age) who weighed <30 kg and >=15 kg at screening starting from Week 4 following a loading dose of 600 mg (2×300 mg injections) on Day 1.
  Interventions: Drug: Dupilumab SAR231893; Drug: non sedating H1-antihistamine
- Study C Placebo (Placebo Comparator): Participants who were omalizumab naïve received placebo matched to dupilumab as SC injection including loading dose from Day 1 up to 24 weeks.
  Interventions: Drug: Placebo; Drug: non sedating H1-antihistamine

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form:Injection solution Route of administration: Subcutaneous
  Arms: Study A Dupilumab; Study B Dupilumab; Study C Dupilumab
Drug: Placebo — Pharmaceutical form:Injection solution Route of administration: Subcutaneous
  Arms: Study A Placebo; Study B Placebo; Study C Placebo
Drug: non sedating H1-antihistamine — Pharmaceutical form:Tablet Route of administration: oral administration

SUMMARY:
Primary Objective:

This study aimed to demonstrate the efficacy of dupilumab in study participants with CSU who remained symptomatic despite the use of H1 antihistamine (Study A and C: omalizumab naïve; Study B: omalizumab intolerant or incomplete responders)

Secondary Objectives:

This study aimed to demonstrate the efficacy of dupilumab on urticaria activity composite endpoint and itch or hives, separately, at various timepoints This study aimed to demonstrate the efficacy of dupilumab on angioedema This study aimed to demonstrate the efficacy of dupilumab on urticaria control This study aimed to demonstrate improvement in health-related quality of life and overall disease status and severity This study aimed to evaluate the ability of dupilumab in reducing the proportion of participants who require treatment with oral corticosteroids (OCS) This study aimed to evaluate safety outcome measures This study aimed to evaluate immunogenicity of dupilumab

DETAILED DESCRIPTION:
The duration of study for each participant included 2-4 weeks of screening period, 24 weeks of treatment period and 12 weeks of post treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Study A and C: Participant were ≥6 years to 80 years of age at the time of signing the informed consent.
* Study B: Participant were ≥12 years (or the minimum legal age for adolescents in the country of the investigational site) to 80 years of age at the time of signing the informed consent
* Participants who had a diagnosis of CSU refractory to H1 antihistamines (H1-AH) at the time of randomization defined by
* Diagnosis of CSU>6 months prior to screening visit
* Presence of itch and hives for >6 consecutive weeks at any time prior to screening visit despite the use of H1-AH during that time period
* Used a study defined H1-antihistamine for CSU treatment
* During the 7 days before randomization:

UAS7≥16 ISS7≥ 8

* Study A and C: omalizumab naïve, Study B; intolerant or incomplete responder to omalizumab
* Participants were willing and able to complete a daily symptom e-Diary for the duration of the study

Exclusion Criteria:

Participants were excluded from any of the studies if any of the following criteria apply:

* Weight was less than 30 kg in adults and adolescents and 15 kg in children aged 6 to<12years
* Clearly defined underlying etiology for chronic urticarias other than CSU
* Presented of skin morbidities other than CSU that may interfere with the assessment of the study outcomes
* Active atopic dermatitis
* Severe concomitant illness(es) that, in the investigator's judgment, would have adversely affected the participant's participation in the study
* Active tuberculosis or non-tuberculous mycobacterial infection, or a history of incompletely treated tuberculosis unless documented adequately treated.
* Diagnosed active endoparasitic infections; suspected or high risk of endoparasitic infection
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiprotozoals, or antifungals within 2 weeks before the screening visit and during the screening period
* Known or suspected immunodeficiency
* Active malignancy or history of malignancy within 5 years before the baseline visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin
* History of systemic hypersensitivity or anaphylaxis to omalizumab or any biologic therapy, including any excipients
* Participation in prior dupilumab clinical study, or have been treated with commercially available dupilumab.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (98):
- United States (16):
  - California Allergy and Asthma Medical Group, Inc. Site Number : 8400019, Los Angeles, California
  - Sarasota Clinical Research Site Number : 8400017, Sarasota, Florida
  - Lenus Research & Medical Group Site Number : 8400001, Sweetwater, Florida
  - University of South Florida Site Number : 8400006, Tampa, Florida
  - Aeroallergy Research Laboratories of Savannah, INC Site Number : 8400018, Savannah, Georgia
  - Allergy & Asthma Specialists, PSC Site Number : 8400020, Owensboro, Kentucky
  - Johns Hopkins University (Asthma and Allergy Center) Site Number : 8400016, Baltimore, Maryland
  - The Clinical Research Center, LLC Site Number : 8400009, St Louis, Missouri
  - UR Dermatology at College Town Site Number : 8400008, Rochester, New York
  - Immunocarolina LLC Site Number : 8400010, Charlotte, North Carolina
  - Bernstein Clinical Research Center Site Number : 8400014, Cincinnati, Ohio
  - Vital Prospects Clinical Research Institute, P.C. Site Number : 8400015, Tulsa, Oklahoma
  - Allergy and Clinical Immunology Associates Site Number : 8400024, Pittsburgh, Pennsylvania
  - National Allergy and ENT Site Number : 8400011, Charleston, South Carolina
  - Pharmaceutical Research & Consulting, Inc. Site Number : 8400003, Dallas, Texas
  - STAAMP Research, LLC Site Number : 8400007, San Antonio, Texas
- Argentina (7):
  - Investigational Site Number : 0320008, CABA, Buenos Aires
  - Investigational Site Number : 0320004, CABA, Buenos Aires
  - Investigational Site Number : 0320006, Rosario, Santa Fe Province
  - Investigational Site Number : 0320007, Rosario, Santa Fe Province
  - Investigational Site Number : 0320005, Rosario, Santa Fe Province
  - Investigational Site Number : 0320003, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320001, Buenos Aires
- Canada (12):
  - Investigational Site Number : 1240009, Calgary, Alberta
  - Investigational Site Number : 1240010, Edmonton, Alberta
  - Investigational Site Number : 1240014, Hamilton, Ontario
  - Investigational Site Number : 1240013, Markham, Ontario
  - Investigational Site Number : 1240003, Niagara Falls, Ontario
  - Investigational Site Number : 1240005, Toronto, Ontario
  - Investigational Site Number : 1240002, Toronto, Ontario
  - Investigational Site Number : 1240007, Windsor, Ontario
  - Investigational Site Number : 1240016, Sherbrooke, Quebec
  - Investigational Site Number : 1240006, Trois-Rivières, Quebec
  - Investigational Site Number : 1240004, Québec
  - Investigational Site Number : 1240011, Québec
- China (9):
  - Investigational Site Number : 1560010, Beijing
  - Investigational Site Number : 1560004, Beijing
  - Investigational Site Number : 1560001, Chengdu
  - Investigational Site Number : 1560007, Guangzhou
  - Investigational Site Number : 1560002, Hangzhou
  - Investigational Site Number : 1560008, Hangzhou
  - Investigational Site Number : 1560006, Jinan
  - Investigational Site Number : 1560003, Shanghai
  - Investigational Site Number : 1560005, Wuxi
- France (8):
  - Investigational Site Number : 2500009, Calais
  - Investigational Site Number : 2500002, Lille
  - Investigational Site Number : 2500011, Mont-de-Marsan
  - Investigational Site Number : 2500004, Nantes
  - Investigational Site Number : 2500012, Nice
  - Investigational Site Number : 2500003, Nice
  - Investigational Site Number : 2500006, Paris
  - Investigational Site Number : 2500005, Pierre-Bénite
- Germany (5):
  - Investigational Site Number : 2760001, Berlin
  - Investigational Site Number : 2760010, Bramsche
  - Investigational Site Number : 2760006, Dresden
  - Investigational Site Number : 2760007, Kiel
  - Investigational Site Number : 2760008, Tübingen
- Hungary (4):
  - Investigational Site Number : 3480005, Debrecen
  - Investigational Site Number : 3480004, Szeged
  - Investigational Site Number : 3480003, Szolnok
  - Investigational Site Number : 3480002, Szombathely
- Japan (12):
  - Investigational Site Number : 3920005, Hiroshima, Hiroshima
  - Investigational Site Number : 3920009, Sapporo, Hokkaido
  - Investigational Site Number : 3920002, Kobe, Hyōgo
  - Investigational Site Number : 3920011, Kagoshima, Kagoshima-ken
  - Investigational Site Number : 3920013, Yokohama, Kanagawa
  - Investigational Site Number : 3920008, Yokohama, Kanagawa
  - Investigational Site Number : 3920003, Suita-shi, Osaka
  - Investigational Site Number : 3920007, Izumo-shi, Shimane
  - Investigational Site Number : 3920006, Itabashi-ku, Tokyo
  - Investigational Site Number : 3920001, Shinagawa-Ku, Tokyo
  - Investigational Site Number : 3920010, Tachikawa-shi, Tokyo
  - Investigational Site Number : 3920004, Nagoya
- Russia (10):
  - Investigational Site Number : 6430008, Chelyabinsk
  - Investigational Site Number : 6430006, Kazan'
  - Investigational Site Number : 6430007, Krasnodar
  - Investigational Site Number : 6430005, Moscow
  - Investigational Site Number : 6430010, Moscow
  - Investigational Site Number : 6430002, Moscow
  - Investigational Site Number : 6430003, Saint Petersburg
  - Investigational Site Number : 6430009, Saratov
  - Investigational Site Number : 6430004, Smolensk
  - Investigational Site Number : 6430001, Stavropol
- Spain (13):
  - Investigational Site Number : 7240012, Santiago de Compostela, A Coruña [La Coruña]
  - Investigational Site Number : 7240003, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240008, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240014, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240010, Esplugues de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number : 7240005, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number : 7240007, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240001, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240006, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240002, Pamplona, Navarre
  - Investigational Site Number : 7240013, Burjassot - Valencia, Valenciana, Comunidad
  - Investigational Site Number : 7240004, Córdoba
  - Investigational Site Number : 7240011, Villarreal de Huerva
- United Kingdom (2):
  - Investigational Site Number : 8260002, London, London, City of
  - Investigational Site Number : 8260001, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Gimenez-Arnau AM, Casale TB, Yosipovitch G, Ensina LF, Inomata N, Msihid J, Makhija M, Radin A, Cyr SL, Sugerman P, Thomas RB, Chuang CC. Dupilumab Improves Health-Related Quality of Life in Omalizumab-Naive Patients with Chronic Spontaneous Urticaria. Dermatol Ther (Heidelb). 2025 Dec 2. doi: 10.1007/s13555-025-01605-w. Online ahead of print. PMID 41326897
- [Derived] Yosipovitch G, Kim BS, Koo JY, Chen Z, Wiggins S, Zahn J, Sugerman P, Haddad EB, Cyr SL. Dupilumab Reduces Pruritus in Clinically Distinct Dermatologic Diseases: Data from Clinical Trials on Atopic Dermatitis, Prurigo Nodularis, and Chronic Spontaneous Urticaria. Dermatol Ther (Heidelb). 2025 Nov 22. doi: 10.1007/s13555-025-01596-8. Online ahead of print. PMID 41272364
- [Derived] Maurer M, Casale TB, Saini SS, Ben-Shoshan M, Laws E, Maloney J, Bauer D, Radin A, Makhija M. Dupilumab Reduces Urticaria Activity, Itch, and Hives in Patients with Chronic Spontaneous Urticaria Regardless of Baseline Serum Immunoglobulin E Levels. Dermatol Ther (Heidelb). 2024 Sep;14(9):2427-2441. doi: 10.1007/s13555-024-01231-y. Epub 2024 Jul 27. PMID 39066978
- See also: EFC16461 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25248&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study comprised of 3 randomized studies of similar design: 2 studies were conducted in participants who were omalizumab naïve (Study A [55 centers in 9 countries] and Study C [50 centers in 9 countries]) and 1 study was conducted in participants who were omalizumab intolerant or incomplete responders (Study B [61 centers in 11 countries]).
Pre-assignment Details: A total of 138 participants in Study A, 108 participants in Study B and 151 participants in Study C were randomized in a 1:1 ratio to receive either weight-tiered dupilumab or matching placebo in respective studies. As pre-specified in the protocol and statistical analysis plan (SAP), the results are presented by study and treatment group/intervention.
Groups:
- Study A: Placebo: Participants who were omalizumab naïve received placebo matched to dupilumab as subcutaneous (SC) injection including loading dose from Day 1 up to 24 weeks.
- Study A: Dupilumab: Participants who were omalizumab naïve received dupilumab for 24 weeks as follows:
  * 300 milligrams (mg) SC injection every 2 weeks (q2w) for adults and those adolescents who weighed >=60 kilograms (kg) at screening starting from Week 2 following a loading dose of 600 mg (2×300 mg injections) on Day 1,
  * 200 mg SC injection q2w for adolescents who weighed <60 kg and children (>=6 to <12 years of age) who weighed >=30 kg at screening starting from Week 2 following a loading dose of 400 mg (2×200 mg injections) on Day 1 and
  * 300 mg SC injection every 4 weeks (q4w) for children (>=6 to <12 years of age) who weighed <30 kg and >=15 kg at screening starting from Week 4 following a loading dose of 600 mg (2×300 mg injections) on Day 1.
- Study B: Placebo: Participants who were intolerant or incomplete responders to omalizumab received placebo matched to dupilumab as SC injection including loading dose from Day 1 up to 24 weeks.
- Study B: Dupilumab: Participants who were intolerant or incomplete responders to omalizumab received dupilumab for 24 weeks as follows:
  * 300 mg SC injection q2w for adults and those adolescents weighing >=60 kg at screening starting from Week 2 following a loading dose of 600 mg (2×300 mg injections) on Day 1 or
  * 200 mg SC injection q2w for adolescents weighing <60 kg at screening starting from Week 2 following a loading dose of 400 mg (2×200 mg injections) on Day 1.
- Study C: Placebo: Participants who were omalizumab naïve received placebo matched to dupilumab as SC injection including loading dose from Day 1 up to 24 weeks.
- Study C: Dupilumab: Participants who were omalizumab naïve received dupilumab for 24 weeks as follows:
  * 300 mg SC injection q2w for adults and those adolescents who weighed >=60 kg at screening starting from Week 2 following a loading dose of 600 mg (2×300 mg injections) on Day 1,
  * 200 mg SC injection q2w for adolescents who weighed <60 kg and children (>=6 to <12 years of age) who weighed >=30 kg at screening starting from Week 2 following a loading dose of 400 mg (2×200 mg injections) on Day 1 and
  * 300 mg SC injection q4w for children (>=6 to <12 years of age) who weighed <30 kg and >=15 kg at screening starting from Week 4 following a loading dose of 600 mg (2×300 mg injections) on Day 1.
Period: Overall Study
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Started | 68 | 70 | 54 | 54 | 77 | 74
Completed | 55 | 63 | 47 | 49 | 67 | 66
Not Completed | 13 | 7 | 7 | 5 | 10 | 8
Not completed — Not related to Coronavirus Disease-2019 (COVID-19) | 2 | 1 | 1 | 3 | 2 | 2
Not completed — Withdrawal by Subject | 8 | 4 | 5 | 2 | 8 | 6
Not completed — Adverse Event | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Poor compliance to protocol | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Study A: Placebo; Study C: Placebo: Participants who were omalizumab naïve received placebo matched to dupilumab as SC injection including loading dose from Day 1 up to 24 weeks.
- Study A: Dupilumab; Study C: Dupilumab: Participants who were omalizumab naïve received dupilumab for 24 weeks as follows:
  * 300 mg SC injection q2w for adults and those adolescents who weighed >=60 kg at screening starting from Week 2 following a loading dose of 600 mg (2×300 mg injections) on Day 1,
  * 200 mg SC injection q2w for adolescents who weighed <60 kg and children (>=6 to <12 years of age) who weighed >=30 kg at screening starting from Week 2 following a loading dose of 400 mg (2×200 mg injections) on Day 1 and
  * 300 mg SC injection q4w for children (>=6 to <12 years of age) who weighed <30 kg and >=15 kg at screening starting from Week 4 following a loading dose of 600 mg (2×300 mg injections) on Day 1.
- Total: Total of all reporting groups
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab | Total
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74 | 397
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (14.8) | 40.7 (16.2) | 46.8 (16.3) | 48.6 (15.6) | 44.0 (16.7) | 45.6 (17.1) | 44.4 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 41 | 41 | 37 | 59 | 47 | 275
  Male | 18 | 29 | 13 | 17 | 18 | 27 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Asian | 16 | 19 | 11 | 6 | 29 | 33 | 114
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 2 | 1 | 2 | 3 | 2 | 0 | 10
  White | 48 | 47 | 41 | 43 | 38 | 32 | 249
  More than one race | 1 | 1 | 0 | 0 | 2 | 1 | 5
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 6 | 7 | 16
Weekly Itch-Severity (ISS7) Score [Mean (Standard Deviation); unit: score on a scale] — ISS was recorded in electronic (e)-diary. The ISS represents severity of itch on a scale ranging from 0 (none) to 3 (intense). The ISS7 score was the sum of daily ISS scores recorded by a participant at the same time each day over 7 days with an overall scale of 0 (no impact) to 21 (severe impact). Higher scores indicated greater intensity of itch. Baseline was defined as the sum of daily scores obtained for 7 days prior to randomization.
  score on a scale | 15.7 (4.1) | 16.1 (4.0) | 16.2 (3.8) | 15.9 (4.0) | 15.0 (3.9) | 15.3 (3.6) | 15.7 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Itch Severity Score at Week 24
Description: ISS was recorded in e-diary. The ISS represents severity of itch on a scale ranging from 0 (none) to 3 (intense). The ISS7 score was the sum of daily ISS scores recorded by a participant at the same time each day over 7 days with an overall scale of 0 (no impact) to 21 (severe impact). Higher scores indicated greater intensity of itch. Least squares (LS) mean is presented. Baseline was defined as the sum of daily scores obtained for 7 days prior to randomization.
Time Frame: Baseline (Day 1) and Week 24
Population: The intent-to-treat (ITT) population included all randomized participants analyzed according to the intervention group allocated by randomization.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
score on a scale | -6.01 (0.94) | -10.24 (0.91) | -4.81 (1.08) | -7.68 (1.10) | -6.10 (1.40) | -8.64 (1.41)
Statistical Analysis 1: Comparison: Study A: Placebo vs Study A: Dupilumab; Analyzed by fitting an analysis of covariance (ANCOVA) model with the corresponding baseline value, intervention group, presence of angioedema at baseline, and regions as covariates; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0005, ANCOVA — Threshold for significance at 2-sided 0.05 level; LS Mean Difference = -4.23, 95% CI 2-sided [-6.63 to -1.84]
Statistical Analysis 2: Comparison: Study B: Placebo vs Study B: Dupilumab; Analyzed by fitting an ANCOVA model with the corresponding baseline value, intervention group, presence of angioedema at baseline, and regions as covariates; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0449, ANCOVA — Threshold for significance at 2-sided 0.043 level; LS Mean Difference = -2.87, 95% CI 2-sided [-5.68 to -0.07]
Statistical Analysis 3: Comparison: Study C: Placebo vs Study C: Dupilumab; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0184, ANCOVA — Threshold for significance at 2-sided 0.05 level; LS Mean Difference = -2.54, 95% CI 2-sided [-4.65 to -0.43]

2. Secondary Outcome: Change From Baseline in Weekly Urticaria Activity Score at Week 24
Description: UAS is a validated composite patient-reported outcome (PRO) measure for assessing chronic spontaneous urticaria (CSU) activity. The once daily UAS is the sum of the daily hives severity score (HSS) and daily ISS recorded in e-diary. Daily HSS assesses number of wheals and range from 0 (none) to 3 (more than 50 hives) whereas daily ISS assesses itch intensity and range from 0 (none) to 3 (intense). The daily UAS scores range from 0 to 6 point/day. Once daily UAS scores are summed over 7-day period to create the UAS7 with an overall scale of 0 (no urticaria) to 42 (severe urticaria). Higher scores indicate greater severity of urticaria symptoms. LS mean is presented. Baseline was defined as the sum of the daily scores for the 7 days prior to the day of randomization.
Time Frame: Baseline (Day 1) and Week 24
Population: The ITT population included all randomized participants analyzed according to the intervention group allocated by randomization.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
score on a scale | -12.00 (1.81) | -20.53 (1.76) | -8.54 (2.14) | -14.37 (2.16) | -11.21 (2.65) | -15.86 (2.66)
Statistical Analysis 1: Comparison: Study A: Placebo vs Study A: Dupilumab; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0003, ANCOVA — Threshold for significance at 2-sided 0.05 level; LS Mean Difference = -8.53, 95% CI 2-sided [-13.16 to -3.90]
Statistical Analysis 2: Comparison: Study C: Placebo vs Study C: Dupilumab; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0226, ANCOVA — Threshold for significance at 2-sided 0.05 level; LS Mean Difference = -4.65, 95% CI 2-sided [-8.65 to -0.65]

3. Secondary Outcome: Change From Baseline in Weekly Hives Severity Score at Week 24
Description: Daily HSS was recorded in e-diary. The HSS7 score is the sum of daily HSS ranging from 0 (none) to 3 (more than 50 hives) recorded by a participant at the same time of each day over 7 days with an overall scale of 0 (no hives) to 21 (severe hives). Higher scores indicate greater intensity of hives. LS mean is presented. Baseline was defined as the sum of the daily scores for the 7 days prior to the day of randomization.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
score on a scale | -5.90 (0.93) | -10.28 (0.91) | -3.63 (1.11) | -6.64 (1.11) | -5.11 (1.31) | -7.27 (1.32)
Statistical Analysis 1: Comparison: Study A: Placebo vs Study A: Dupilumab; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0003, ANCOVA — Threshold for significance at 2-sided 0.05 level; LS Mean Difference = -4.38, 95% CI 2-sided [-6.78 to -1.98]
Statistical Analysis 2: Comparison: Study C: Placebo vs Study C: Dupilumab; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0316, ANCOVA — Threshold for significance at 2-sided 0.05 level; LS Mean Difference = -2.17, 95% CI 2-sided [-4.15 to -0.19]

4. Secondary Outcome: Percentage of Responders for Weekly Itch Severity Score Minimally Important Difference (MID) at Week 24
Description: The ISS represents severity of itch on a scale ranging from 0 (none) to 3 (intense). The ISS7 score was the sum of daily ISS scores recorded by a participant at the same time each day over 7 days with an overall scale of 0 (no impact) to 21 (severe impact). Higher scores indicated greater intensity of itch. An ISS7 MID response was defined as >=5 points decrease from baseline after study intervention.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
percentage of participants | 42.6 | 72.9 | 38.9 | 59.3 | 51.9 | 70.3
Statistical Analysis 1: Comparison: Study A: Placebo vs Study A: Dupilumab; Cochran-Mantel-Haenszel (CMH) test was performed on association between responder status and intervention group, adjusted by baseline disease severity (UAS7<28,>=28), presence of angioedema at baseline and region; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0014, Cochran-Mantel-Haenszel — Threshold for significance at 2-sided 0.05 level; Odds Ratio (OR) = 3.413, 95% CI 2-sided [1.596 to 7.299]
Statistical Analysis 2: Comparison: Study C: Placebo vs Study C: Dupilumab; CMH test was performed on the association between the responder status and intervention group, adjusted by baseline disease severity (UAS7 <28, >=28), presence of angioedema at baseline, and region; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0109, Cochran-Mantel-Haenszel — Threshold for significance at 2-sided 0.05 level; Odds Ratio (OR) = 2.507, 95% CI 2-sided [1.231 to 5.107]

5. Secondary Outcome: Percentage of Participants With Weekly Urticaria Activity Score <=6 at Week 24
Description: UAS is a validated composite PRO measure for assessing CSU activity. The once daily UAS is the sum of the daily HSS and daily ISS recorded in e-diary. Daily HSS assesses number of wheals and range from 0 (none) to 3 (more than 50 hives) whereas daily ISS assesses itch intensity and range from 0 (none) to 3 (intense). The daily UAS scores range from 0 to 6 point/day. Once daily UAS scores are summed over 7-day period to create the UAS7 with an overall scale of 0 (no urticaria) to 42 (severe urticaria). Higher scores indicate greater severity of urticaria symptoms. In evaluating urticaria control using UAS7, an UAS7 score of <=6 indicated a well-controlled urticaria.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
percentage of participants | 23.5 | 45.7 | 18.5 | 24.1 | 23.4 | 40.5
Statistical Analysis 1: Comparison: Study A: Placebo vs Study A: Dupilumab; [analysis description as in outcome 4, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0075, Cochran-Mantel-Haenszel — Threshold for significance at 2-sided 0.05 level; Odds Ratio (OR) = 2.848, 95% CI 2-sided [1.301 to 6.234]
Statistical Analysis 2: Comparison: Study C: Placebo vs Study C: Dupilumab; [analysis description as in outcome 4, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0045, Cochran-Mantel-Haenszel — Threshold for significance at 2-sided 0.05 level; Odds Ratio (OR) = 3.137, 95% CI 2-sided [1.371 to 7.176]

6. Secondary Outcome: Percentage of Participants With Weekly Urticaria Activity Score =0 at Week 24
Description: UAS is a validated composite PRO measure for assessing CSU activity. The once daily UAS is the sum of the daily HSS and daily ISS recorded in e-diary. Daily HSS assesses number of wheals and range from 0 (none) to 3 (more than 50 hives) whereas daily ISS assesses itch intensity and range from 0 (none) to 3 (intense). The daily UAS scores range from 0 to 6 point/day. Once daily UAS scores are summed over 7-day period to create the UAS7 with an overall scale of 0 (no urticaria) to 42 (severe urticaria). Higher scores indicate greater severity of urticaria symptoms. In evaluating urticaria control using UAS7, an UAS7 score of 0 indicated an absence of both itch and hives and a complete resolution of CSU symptoms.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
percentage of participants | 13.2 | 31.4 | 9.3 | 13.0 | 18.2 | 29.7
Statistical Analysis 1: Comparison: Study A: Placebo vs Study A: Dupilumab; [analysis description as in outcome 4, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0199, Cochran-Mantel-Haenszel — Threshold for significance at 2-sided 0.05 level; Odds Ratio (OR) = 2.908, 95% CI 2-sided [1.173 to 7.209]
Statistical Analysis 2: Comparison: Study C: Placebo vs Study C: Dupilumab; [analysis description as in outcome 4, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0187, Cochran-Mantel-Haenszel — Threshold for significance at 2-sided 0.05 level; Odds Ratio (OR) = 2.677, 95% CI 2-sided [1.127 to 6.359]

7. Secondary Outcome: Change From Baseline in Urticaria Control Test (UCT) at Week 24
Description: The UCT assessed urticaria control based on 4 items (severity of pruritus and wheals urticaria symptoms; frequency of treatment being not sufficient; quality-of-life [QoL] impairment; overall urticarial control). Each item was rated on a 5-point Likert-type scale from 0 (no control) to 4 (maximum control). The overall UCT score was the sum of all 4 individual item scores with a range of 0 (no disease control) to 16 (complete disease control). Higher scores indicated greater disease control. LS mean is presented. Baseline was defined as the last available value up to randomization date and prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
score on a scale | 4.88 (0.61) | 7.71 (0.59) | 3.38 (0.74) | 5.33 (0.77) | 4.16 (0.94) | 5.09 (0.95)
Statistical Analysis 1: Comparison: Study C: Placebo vs Study C: Dupilumab; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.1940, ANCOVA — Threshold for significance at 2-sided 0.05 level; LS Mean Difference = 0.93, 95% CI 2-sided [-0.48 to 2.34]

8. Secondary Outcome: Change From Baseline in Weekly Itch Severity Score at Week 12
Description: ISS was recorded in e-diary. The ISS represents severity of itch on a scale ranging from 0 (none) to 3 (intense). The ISS7 score was the sum of daily ISS scores recorded by a participant at the same time each day over 7 days with an overall scale of 0 (no impact) to 21 (severe impact). Higher scores indicated greater intensity of itch. LS mean is presented. Baseline was defined as the sum of daily scores obtained for 7 days prior to randomization.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
score on a scale | -6.01 (0.85) | -8.37 (0.84) | -4.52 (0.95) | -7.37 (0.97) | -5.31 (1.32) | -7.15 (1.32)
Statistical Analysis 1: Comparison: Study A: Placebo vs Study A: Dupilumab; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0377, ANCOVA — Threshold for significance at 2-sided 0.05 level; LS Mean Difference = -2.37, 95% CI 2-sided [-4.60 to -0.13]

9. Secondary Outcome: Change From Baseline in Weekly Urticaria Activity Score at Week 12
Description: UAS is a validated composite PRO measure for assessing CSU activity. The once daily UAS is the sum of the daily HSS and daily ISS recorded in e-diary. Daily HSS assesses number of wheals and range from 0 (none) to 3 (more than 50 hives) whereas daily ISS assesses itch intensity and range from 0 (none) to 3 (intense). The daily UAS scores range from 0 to 6 point/day. Once daily UAS scores are summed over 7-day period to create the UAS7 with an overall scale of 0 (no urticaria) to 42 (severe urticaria). Higher scores indicate greater severity of urticaria symptoms. LS mean is presented. Baseline was defined as the sum of the daily scores for the 7 days prior to the day of randomization.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
score on a scale | -11.79 (1.64) | -16.81 (1.62) | -8.22 (1.91) | -13.33 (1.94) | -9.51 (2.54) | -12.87 (2.54)
Statistical Analysis 1: Comparison: Study A: Placebo vs Study A: Dupilumab; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0223, ANCOVA — Threshold for significance at 2-sided 0.05 level; LS Mean Difference = -5.02, 95% CI 2-sided [-9.32 to -0.72]

10. Secondary Outcome: Percentage of Participants With Weekly Urticaria Activity Score <=6 and =0 at Week 12
Description: UAS is a validated composite PRO measure for assessing CSU activity. The once daily UAS is the sum of the daily HSS and daily ISS recorded in e-diary. Daily HSS assesses number of wheals and range from 0 (none) to 3 (more than 50 hives) whereas daily ISS assesses itch intensity and range from 0 (none) to 3 (intense). The daily UAS scores range from 0 to 6 point/day. Once daily UAS scores are summed over 7-day period to create the UAS7 with an overall scale of 0 (no urticaria) to 42 (severe urticaria). Higher scores indicate greater severity of urticaria symptoms. In evaluating urticaria control using UAS7, an UAS7 score of <=6 indicated a well-controlled urticaria and an UAS7 score of 0 indicated an absence of both itch and hives and a complete resolution of CSU symptoms.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
percentage of participants
  UAS7 <=6 | 17.6 | 34.3 | 9.3 | 24.1 | 16.9 | 31.1
  UAS7=0 | 8.8 | 15.7 | 1.9 | 13.0 | 11.7 | 17.6
Statistical Analysis 1: Comparison: Study A: Placebo vs Study A: Dupilumab; [analysis description as in outcome 4, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0215, Cochran-Mantel-Haenszel — Threshold for significance at 2-sided 0.05 level; Odds Ratio (OR) = 2.645, 95% CI 2-sided [1.154 to 6.061]

11. Secondary Outcome: Percentage of Responders for Weekly Itch Severity Score Minimally Important Difference at Week 12
Description: as for outcome 4
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
percentage of participants | 52.9 | 70.0 | 46.3 | 64.8 | 51.9 | 58.1
Statistical Analysis 1: Comparison: Study A: Placebo vs Study A: Dupilumab; [analysis description as in outcome 4, analysis 2]; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error; p = 0.0971, Cochran-Mantel-Haenszel — Threshold for significance at 2-sided 0.05 level; Odds Ratio (OR) = 1.872, 95% CI 2-sided [0.893 to 3.923]

12. Secondary Outcome: Change From Baseline in Weekly Hives Severity Score at Week 12
Description: as for outcome 3
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
score on a scale | -5.69 (0.83) | -8.39 (0.83) | -3.71 (1.01) | -5.97 (1.02) | -4.22 (1.28) | -5.75 (1.28)

13. Secondary Outcome: Change From Baseline in Urticaria Control Test at Week 12
Description: as for outcome 7
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
score on a scale | 4.62 (0.57) | 6.48 (0.57) | 3.11 (0.65) | 5.48 (0.67) | 3.26 (0.88) | 4.61 (0.89)

14. Secondary Outcome: Change From Baseline in Weekly Itch Severity Score at Weeks 4, 8, 16 and 20
Description: ISS was recorded in e-diary. The ISS represents severity of itch on a scale ranging from 0 (none) to 3 (intense). The ISS7 score was the sum of daily ISS scores recorded by a participant at the same time each day over 7 days with an overall scale of 0 (no impact) to 21 (severe impact). Higher scores indicated greater intensity of itch. Mean is presented. Baseline was defined as the sum of daily scores obtained for 7 days prior to randomization.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16 and 20
Population: The ITT population included all randomized participants analyzed according to the intervention group allocated by randomization. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 65 | 70 | 54 | 54 | 72 | 70
score on a scale
  Week 4: number analyzed (Participants) | 65 | 70 | 54 | 54 | 72 | 69
  Week 4 | -3.30 (6.54) | -4.96 (5.49) | -4.12 (6.28) | -5.51 (5.64) | -3.78 (4.73) | -5.26 (5.16)
  Week 8: number analyzed (Participants) | 62 | 68 | 50 | 52 | 70 | 69
  Week 8 | -4.98 (7.49) | -6.99 (6.78) | -4.27 (5.92) | -7.25 (6.29) | -4.92 (5.67) | -7.83 (6.02)
  Week 16: number analyzed (Participants) | 58 | 66 | 50 | 51 | 68 | 70
  Week 16 | -5.61 (7.45) | -9.43 (6.86) | -4.52 (6.68) | -8.05 (7.43) | -6.22 (5.78) | -8.24 (7.37)
  Week 20: number analyzed (Participants) | 57 | 64 | 49 | 50 | 67 | 66
  Week 20 | -6.40 (7.82) | -10.04 (7.22) | -5.35 (7.17) | -7.54 (7.94) | -6.64 (6.43) | -9.27 (6.58)

15. Secondary Outcome: Time to First Weekly Itch Severity Score Minimally Important Difference Response During the 24-Week Treatment Period
Description: The ISS represents severity of itch on a scale ranging from 0 (none) to 3 (intense). The ISS7 score was the sum of daily ISS scores recorded by a participant at the same time each day over 7 days with an overall scale of 0 (no impact) to 21 (severe impact). Higher scores indicated greater intensity of itch. The MID for ISS7 was a change of 5.0 points. Time to first ISS7 MID response (ISS7 >=5) was defined as time to reduction from baseline of 5 points or more. Kaplan-Meier estimate is presented. Baseline was defined as the sum of daily scores obtained for 7 days prior to randomization.
Time Frame: Baseline (Day 1) up to Week 24
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
weeks | 4.0 [2.0 to 8.0] | 3.0 [2.0 to 5.0] | 4.0 [2.0 to 7.0] | 3.0 [2.0 to 4.0] | 5.0 [3.0 to 7.0] | 3.5 [3.0 to 5.0]

16. Secondary Outcome: Change From Baseline in Angioedema Activity Score Over 7 Days (AAS7) at Weeks 12 and 24
Description: The AAS is a diary in which participants document on a daily basis the presence or absence of angioedema during the past 24 hours. If angioedema is present, participants answer 5 additional questions about the time of the day the swelling episode occurred and the severity and impact on daily functioning and appearance this swelling episode has had. Each AAS item is scored between 0 (minimum) and 3 (maximum). The daily AASs range from 0 (no episode) to 15 (severe) points. The AAS7 score is the sum of daily AAS scores reported by a participant at the same time of each day over 7 days, with a range of 0 (no angioedema episodes) to 105 (highest angioedema severity). Higher scores indicate greater angioedema activity. Mean is presented. Baseline was defined as the sum of the daily scores for the 7 days prior to the day of randomization.
Time Frame: Baseline (Day 1) and Weeks 12 and 24
Population: The ITT population included all randomized participants analyzed according to the intervention group allocated by randomization. Only those participants with angioedema at baseline and with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 31 | 27 | 32 | 20 | 21 | 12
score on a scale
  Week 12: number analyzed (Participants) | 31 | 27 | 32 | 19 | 18 | 11
  Week 12 | -23.46 (21.76) | -19.14 (18.89) | -16.74 (21.74) | -19.41 (34.44) | -32.14 (32.15) | -34.33 (36.19)
  Week 24: number analyzed (Participants) | 29 | 26 | 28 | 20 | 21 | 12
  Week 24 | -23.56 (23.04) | -18.76 (22.85) | -15.83 (25.73) | -13.95 (37.22) | -31.00 (36.38) | -36.28 (27.61)

17. Secondary Outcome: Percentage of Well-controlled Participants (Urticaria Control Test >=12) at Weeks 12 and 24
Description: The UCT assessed urticaria control based on 4 items (severity of pruritus and wheals urticaria symptoms; frequency of treatment being not sufficient; QoL impairment; overall urticarial control). Each item was rated on a 5-point Likert-type scale from 0 (no control) to 4 (maximum control). The overall UCT score was the sum of all 4 individual item scores with a range of 0 (no disease control) to 16 (complete disease control). Higher scores indicated greater disease control. An UCT score of >=12 (out of maximum 16) indicated a well-controlled urticaria disease status.
Time Frame: Weeks 12 and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
percentage of participants
  Week 12 | 27.9 | 44.3 | 18.5 | 51.9 | 22.1 | 37.8
  Week 24 | 30.9 | 48.6 | 20.4 | 44.4 | 39.0 | 50.0

18. Secondary Outcome: Change From Baseline in Health-related Quality-of-life (HRQoL) as Measured by Dermatology Life Quality Index (DLQI) in Participants >=16 Years Old at Weeks 12 and 24
Description: The DLQI is an assessment assessing the impact of skin disease on participants' HRQoL over the previous week and contains 10 questions related to symptoms, leisure activities, work/school or holiday time, personal relationships including intimate, the side effects of treatment, and emotional reactions to having a skin disease. The questions (except question 7) were scored on a 4-point Likert scale: 0 (not at all), 1 (a little), 2 (a lot), 3 (very much). Question 7 about work/studying asked whether work/study had been prevented and then (if "No") to what degree the skin condition has been a problem at work/study; the item was again rated on a 3-point Likert scale: 0 (not at all) to 3 (a lot). Total DLQI was calculated by summing the score of each question and ranged from 0 (no impact) to 30 (severe impact). Higher scores indicated poor HRQoL. Mean is presented. Baseline was defined as the last available value up to randomization date and prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) and Weeks 12 and 24
Population: The ITT population included all randomized participants analyzed according to the intervention group allocated by randomization. Only those participants >=16 years with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 65 | 65 | 51 | 47 | 67 | 70
score on a scale
  Week 12 | -7.55 (7.47) | -8.55 (6.27) | -4.53 (6.28) | -6.77 (6.92) | -5.01 (6.25) | -6.61 (7.04)
  Week 24: number analyzed (Participants) | 61 | 64 | 49 | 45 | 63 | 67
  Week 24 | -7.56 (8.13) | -9.50 (5.92) | -4.96 (6.87) | -6.91 (7.51) | -6.81 (6.54) | -8.09 (7.66)

19. Secondary Outcome: Change From Baseline in Health-related Quality-of-life as Measured by Children's Dermatology Life Quality Index (CDLQI) in Participants >=6 to <16 Years Old at Weeks 12 and 24
Description: The CDLQI is a validated questionnaire designed to measure the impact of skin disease on children's HRQoL. Participants provide responses to 10 questions (symptoms feelings associated with disease, the impact of the disease on leisure, school or holidays, personal relationships, sleep, and side effects of treatment for the skin disease). The instrument has a recall period of 7 days. 9 of the 10 questions are scored on a 4-point Likert scale ranging from 0 (not at all/question unanswered) to 3 (very much). Question 7 has an additional possible response (prevented school) which is assigned a score of 3 (0 [not at all] to 3 [definitely]). The total CDLQI score is the sum of the score of each question ranging 0 (no impact) to 30 (severe impact). The higher the score, the greater the impact is on the child's HRQoL. Mean is presented. Baseline was defined as the last available value up to randomization date and prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) and Weeks 12 and 24
Population: The ITT population included all randomized participants analyzed according to the intervention group allocated by randomization. Only those participants >=6 and <16 years with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 1 | 2 | 0 | 1 | 5 | 2
score on a scale
  Week 12 | -5.00 (NA) — NA indicates that standard deviation could not be calculated for 1 participant. | -8.00 (5.66) |  | -7 (NA) — NA indicates that standard deviation could not be calculated for 1 participant. | -4.60 (10.04) | -9.00 (2.83)
  Week 24: number analyzed (Participants) | 0 | 2 | 0 | 1 | 5 | 2
  Week 24 |  | -12.50 (12.02) |  | -7 (NA) — NA indicates that standard deviation could not be calculated for 1 participant. | -5.60 (7.83) | -4.50 (7.78)

20. Secondary Outcome: Patient Global Impression of Change (PGIC) of Chronic Spontaneous Urticaria at Weeks 12 and 24
Description: The PGIC is a 1-item questionnaire that asks the participant to provide the overall self-assessment of change in their CSU on a 7-point scale compared to just before participant started taking the study intervention. Response choices are: 0 (very much better), 1 (moderately better), 2 (a little better), 3 (no change), 4 (a little worse), 5 (moderately worse), 6 (very much worse). Higher score indicate worsening.
Time Frame: Weeks 12 and 24
Population: The ITT population included all randomized participants analyzed according to the intervention group allocated by randomization. Only those participants with data collected at Weeks 12 and 24 are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 66 | 69 | 54 | 52 | 73 | 73
score on a scale
  Week 12 | 1.68 (1.43) | 1.10 (1.24) | 2.06 (1.29) | 1.62 (1.46) | 1.59 (1.23) | 1.27 (1.44)
  Week 24: number analyzed (Participants) | 61 | 68 | 50 | 50 | 68 | 70
  Week 24 | 1.70 (1.50) | 1.04 (1.51) | 1.90 (1.64) | 1.44 (1.55) | 1.18 (1.36) | 1.01 (1.48)

21. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity (PGIS) of Chronic Spontaneous Urticaria at Weeks 12 and 24
Description: The PGIS is a 1-item questionnaire that asks participants to provide the overall self-assessment of their disease severity on a 4-point scale for the past week. Response choices are: 1 (none), 2 (mild), 3 (moderate), 4 (severe). Higher score indicate more severity. Baseline was defined as the last available value up to randomization date and prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) and Weeks 12 and 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 66 | 69 | 54 | 52 | 73 | 73
score on a scale
  Week 12 | -0.89 (0.98) | -1.23 (0.93) | -0.46 (0.93) | -1.15 (1.04) | -0.82 (0.98) | -0.95 (0.97)
  Week 24: number analyzed (Participants) | 61 | 68 | 50 | 50 | 68 | 70
  Week 24 | -0.97 (1.18) | -1.44 (0.92) | -0.54 (1.16) | -0.96 (1.05) | -1.03 (1.09) | -1.33 (1.05)

22. Secondary Outcome: Time to First Oral Corticosteroid (OCS) Use for Chronic Spontaneous Urticaria During the 24-week Treatment Period
Description: Participants receiving OCS as rescue medications for CSU were recorded by the Investigator in e-case report form (eCRF) during the 24-week treatment period. Kaplan-Meier estimate for time to first OCS use is presented.
Time Frame: Baseline (Day 1) up to Week 24
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
weeks | 0.110 [0.048 to 0.200] | 0.087 [0.035 to 0.168] | 0.158 [0.074 to 0.271] | 0.116 [0.047 to 0.220] | 0.067 [0.025 to 0.138] | 0.014 [0.001 to 0.068]

23. Secondary Outcome: Percentage of Participants Receiving Oral Corticosteroid for Chronic Spontaneous Urticaria During the 24-week Treatment Period
Description: Percentage of participants receiving OCS as rescue medications for CSU were recorded by the Investigator in eCRF during the 24-week treatment period.
Time Frame: Baseline (Day 1) up to Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
percentage of participants | 10.3 | 8.6 | 14.8 | 11.1 | 6.5 | 1.4

24. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were defined as AEs that developed, worsened or became serious during the TE period.
Time Frame: From first dose of study intervention (Day 1) up to end of follow-up, approximately 36 weeks each for Study A, B and C
Population: The safety population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. As pre-specified in the protocol and SAP, the results are presented by study and treatment group/intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 68 | 70 | 54 | 54 | 77 | 74
Participants
  TEAEs | 40 | 38 | 29 | 33 | 41 | 40
  TESAEs | 5 | 2 | 2 | 3 | 1 | 5

25. Secondary Outcome: Number of Participants With Treatment-emergent Anti-drug Antibodies (ADA) Against Dupilumab
Description: Blood samples were collected at specified timepoints and ADA samples were assayed using validated methods. Treatment-emergent ADA response was defined as a positive response in the ADA assay post first dose when baseline results were negative or missing. Number of participants with treatment-emergent ADA response is presented.
Time Frame: Up to Week 24
Population: The ADA population included all participants in the safety population who had at least 1 non-missing ADA result after first dose of the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
Number analyzed (Participants) | 66 | 69 | 53 | 52 | 75 | 72
Participants | 1 | 9 | 2 | 10 | 0 | 1

ADVERSE EVENTS:
Time Frame: From first dose of study intervention (Day 1) up to end of follow-up, approximately 36 weeks each for Study A, B and C
Description: Analysis was performed on the safety population. As pre-specified in the protocol and SAP, the results are presented by study and treatment group/intervention.
Arm/Group | Study A: Placebo | Study A: Dupilumab | Study B: Placebo | Study B: Dupilumab | Study C: Placebo | Study C: Dupilumab
All-Cause Mortality (participants affected / at risk) | 1/68 | 0/70 | 0/54 | 0/54 | 0/77 | 0/74
Serious Adverse Events (participants affected / at risk) | 5/68 | 2/70 | 2/54 | 3/54 | 1/77 | 5/74
Other Adverse Events (participants affected / at risk) | 19/68 | 12/70 | 15/54 | 17/54 | 15/77 | 20/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study A: Placebo (N=68) | Study A: Dupilumab (N=70) | Study B: Placebo (N=54) | Study B: Dupilumab (N=54) | Study C: Placebo (N=77) | Study C: Dupilumab (N=74)
Covid-19 Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed Suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic Spontaneous Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study A: Placebo (N=68) | Study A: Dupilumab (N=70) | Study B: Placebo (N=54) | Study B: Dupilumab (N=54) | Study C: Placebo (N=77) | Study C: Dupilumab (N=74)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1) | 4 (4) | 5 (5) | 4 (4) | 6 (6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 4 (5) | 1 (1) | 6 (6) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Chronic Spontaneous Urticaria (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (4) | 3 (4) | 6 (8) | 3 (4) | 2 (2)
Injection Site Erythema (General disorders) | 4 (9) | 3 (13) | 3 (4) | 0 (0) | 0 (0) | 4 (10)
Injection Site Reaction (General disorders) | 2 (10) | 4 (9) | 1 (2) | 1 (1) | 1 (1) | 3 (8)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT04180488/Prot_002.pdf
  • Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT04180488/SAP_003.pdf